CLINICAL TRIAL: NCT05455658
Title: A Phase II Trial of The Immunogenicity of a DNA Plasmid Based Vaccine (STEMVAC) Encoding Th1 Selective Epitopes From Five Antigens Associated With Breast Cancer Stem Cells (MDM2, YB1, SOX2, CDC25B, CD105) in Participants With Early Stage Triple Negative Breast Cancer
Brief Title: STEMVAC in Patients With Early Stage Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1122380; NCI-2021-07734 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UG1CA242635 (NIH); UWI20-00-01 (Other: DCP Identifier)
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (STEMVAC vaccine, sargramostim) (Experimental): Patients receive STEMVAC vaccine with sargramostim ID every month for 3 months in the absence of disease progression or unacceptable toxicity. Patients then receive STEMVAC vaccine with sargramostim ID booster injections 3 months after the 3rd vaccination and 6 months after the 1st booster vaccination.
  Interventions: Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine; Biological: Sargramostim

INTERVENTIONS:
Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine — Given IV
  Other Names: CD105/Yb-1/SOX2/CDH3/MDM2 Plasmid Vaccine; STEMVAC; STEMVAC Th1 Polyepitope Plasmid-based Vaccine
Biological: Sargramostim — Given ID
  Other Names: 123774-72-1; 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase II trial studies the effect of DNA plasmid based vaccine (STEMVAC) in treating patients with patients with stage IB-III triple negative breast cancer. STEMVAC may wake up the immune system in patients who have had a diagnosis of triple negative breast cancer and have been treated. STEMVAC targets proteins that are expressed on breast cancer cells and works by boosting the immune system to recognize and destroy the invader cancer cell proteins that are causing the disease. The purpose of this trial is to test the immune system's response to STEMVAC.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive STEMVAC vaccine with sargramostim intradermally (ID) every month for 3 months in the absence of disease progression or unacceptable toxicity. Patients then receive STEMVAC vaccine with sargramostim ID booster injections 3 months after the 3rd vaccination and 6 months after the 1st booster vaccination.

After completion of study treatment, patients are followed up at 28 days, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with triple negative breast cancer, stages IB, II or III. Estrogen receptor (ER)-negative and progesterone receptor (PR)-negative is defined as breast cancer with less than 10% of ER or PR expression. HER2 negative is defined as:

  * 0-1+ HER2 expression by immunohistochemistry (IHC) OR
  * Fluorescence in situ hybridization (FISH) negative OR
  * HER2 2+ and FISH negative
  * Note: Participants with low ER positivity (≤10%) who are already on adjuvant hormonal therapy will be allowed on study and can continue their adjuvant hormonal treatment during study participation.
* Participants must have completed all standard of care (or investigational) systemic therapy (including immune modulating agents) and radiotherapy if used between 28 and 365 days prior to enrollment

  * Note: Treatment with a bisphosphonate or denosumab to prevent bone loss is not considered to be systemic therapy for breast cancer and its use within the 28 day pre-enrollment period or while on study is not exclusionary. Treatment with adjuvant olaparib within the 28 day pre-enrollment period or while on study is not exclusionary.
* Participants must agree to avoid systemic steroids for the duration of the treatment period and until completion of the 1 month post 2nd booster vaccine visit (end of treatment)
* Participants must be at least 18 years of age

  * Note: Because no dosing or adverse event (AE) data are currently available on the use of STEMVAC in participants < 18 years of age, children and adolescents are excluded from this study but will be eligible for future pediatric trials, if applicable.
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1
* White blood cell (WBC) >= 3000/mm^3 (within 60 days of enrollment and at least 28 days post standard of care [SOC] treatment)
* Lymphocyte count >= 800/mm^3 (within 60 days of enrollment and at least 28 days post standard of care [SOC] treatment)
* Platelet count >= 100,000/mm^3 (within 60 days of enrollment and at least 28 days post standard of care [SOC] treatment)
* Hemoglobin (Hgb) >= 10 g/dl (within 60 days of enrollment and at least 28 days post standard of care [SOC] treatment)
* Serum creatinine =< 1.2 mg/dl OR creatinine clearance > 60 ml/min (within 60 days of enrollment and at least 28 days post standard of care [SOC] treatment)
* Total bilirubin =< 1.5 X upper limit of institutional normal (ULN) (within 60 days of enrollment and at least 28 days post standard of care [SOC] treatment)
* AST (aspartate aminotransferase)/serum glutamic-oxaloacetic transaminase (SGOT) =< 1.5 X upper limit of institutional normal (ULN) (within 60 days of enrollment and at least 28 days post standard of care [SOC] treatment)
* Must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator, not have any significant active concurrent medical illnesses or condition precluding protocol treatment
* The effects of STEMVAC on the developing human fetus are unknown. For this reason,

  * Female participant agrees to use adequate contraception (examples include: estrogen and/or progestogen containing hormonal contraception, barrier method (condom, cervical cap) or abstinence) while on the study and until 1 month after the 2nd booster vaccination when/if engaging in sex that could lead to pregnancy. Exceptions: Females who have had a hysterectomy, tubal ligation or bilateral oophorectomy OR meet one of the following criteria for postmenopausal: Age > 60 or age < 60 with >= 12 months amenorrhea and follicle-stimulating hormone (FSH) within the testing facility's postmenopausal range
  * Female participant agrees to inform her study physician immediately should she become pregnant or suspect she is pregnant while participating in this study
  * Male participants who are having sex that can lead to pregnancy must use an acceptable form of contraception (vasectomy with the absence of sperm, sexual abstinence, condoms) throughout the course of the study
  * Must be 14 days between a vaccine (i.e. COVID19, Flu, shingrix, Tdap, etc.) and any STEMVAC vaccination. **Note: This does not apply to the Td vaccine.
* Patients must be willing to not undergo major elective surgical procedures with general anesthesia or conscious sedation through the end of treatment visit. (Note: port removal is allowable)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Contraindication or known hypersensitivity to receiving sargramostim (rhuGM-CSF) or other products
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to STEMVAC
* Participants receiving any other investigational agents
* Chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs) is prohibited during the treatment period of the study, except when taken as low-dose (81 mg) aspirin therapy. Prohibited chronic use is defined as daily use for more than 7 days
* Participants with any clinically significant autoimmune disease uncontrolled with treatment
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women are excluded from this study
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C

  * Note: These individuals are excluded in order to avoid confounding an existing condition with an immune response to STEMVAC
* Chronic usage of immunosuppressants and glucocorticoids (methotrexate for RA, etc.)
* History of invasive breast cancer prior to TNBC diagnosis * Note: Prior DCIS is allowable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2028-07-16 (Estimated)

PRIMARY OUTCOMES:
Cellular immune response: incidence | At 1 month after 3rd vaccination
  Defined by the incidence of development of the Th1 (IFN-gamma [g]) antigen specific immune response against STEMVAC antigens using enzyme-linked immunosorbent spot assay (ELISPOT).
Cellular immune response: incidence | At 10 months after 3rd vaccination
  Defined by the incidence of development of the Th1 (IFN-gamma [g]) antigen specific immune response against STEMVAC antigens using enzyme-linked immunosorbent spot assay (ELISPOT).
Cellular immune response: magnitude | At 1 month after 3rd vaccination
  Defined by the magnitude of development of the Th1 (IFN-gamma [g]) antigen specific immune response against STEMVAC antigens using enzyme-linked immunosorbent spot assay (ELISPOT). The magnitude of immune response is defined as the sum of the corrected spots/well values calculated at each time point.
Cellular immune response: magnitude | At 3 months after 3rd vaccination
  Defined by the magnitude of development of the Th1 (IFN-gamma [g]) antigen specific immune response against STEMVAC antigens using enzyme-linked immunosorbent spot assay (ELISPOT). The magnitude of immune response is defined as the sum of the corrected spots/well values calculated at each time point.
Cellular immune response: magnitude | At 9 months after 3rd vaccination
  Defined by the magnitude of development of the Th1 (IFN-gamma [g]) antigen specific immune response against STEMVAC antigens using enzyme-linked immunosorbent spot assay (ELISPOT). The magnitude of immune response is defined as the sum of the corrected spots/well values calculated at each time point.
Cellular immune response: magnitude | At 10 months after 3rd vaccination
  Defined by the magnitude of development of the Th1 (IFN-gamma [g]) antigen specific immune response against STEMVAC antigens using enzyme-linked immunosorbent spot assay (ELISPOT). The magnitude of immune response is defined as the sum of the corrected spots/well values calculated at each time point.

SECONDARY OUTCOMES:
Kinetics of the magnitude of antigen specific IFN-gamma ELISPOT counts | 13 months
  Will be assessed over time from pre to post immunization to determine if pre-existent immunity affects magnitude of response.
Incidence of adverse events | 1 month after last booster vaccine
  Safety and systemic toxicity will be determined by chemical and clinical parameters evaluated at various time points. Toxicity grading will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 and monitoring of adverse events will be done per Food and Drug Administration and NCI guidelines.
Activation status and repertoire diversity of peripheral blood T-cells | Prior to and after STEMVAC vaccination
  The peripheral T cell repertoire diversity will be determined by high-throughput deoxyribonucleic acid (DNA) sequencing of the recombined V(D)J region of the T cell receptor beta-chain (TCRB) using the immunoSEQ platform (Adaptive Biotechnologies) on antigen-specific T-cells from a short-term in vitro culture. The activation, exhaustion and memory status of the peripheral T cells will be determined by flow cytometry using fluorochrome linked antibodies to PD-1, CD4, CD3, LAG3, CD137, CD8, KLGR1, CD44, CD69, CD62L and OX40. Transcription factors for Th1 (Tbet), Th2 (GATA3) and Treg (FOXP3) will also be evaluated. All results will be summarized using simple descriptive statistics.
Relapse free survival (RFS) | Up to 5 years
  Will explore if adjuvant vaccination with STEMVAC improves relapse free survival as compared to historical controls. Local and distant recurrence at year 5 will be reported as proportion with confidence intervals, and RFS will be estimated using Kaplan-Meier method with the 5-year RFS rate estimated from the Kaplan-Meier estimate of the survival distribution along with a 95% confidence interval. Comparison of the local and distant recurrence and 5-year RFS against the historical control will be based on a binomial test.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Disis, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Howard Bailey, MD, Study Director — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05455658/ICF_000.pdf